CLINICAL TRIAL: NCT01018225
Title: Exploratory Study Evaluating the Effects of Darifenacin on Nocturia, Sleep and Daytime Wakefulness
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was cancelled due to lack of enrollment
Sponsor: Cognitive Research Corporation (Industry)
Collaborators: Novartis Pharmaceuticals (Industry)
Other Study IDs: CRC090001
Record Dates: First submitted 2009-11-20; First posted 2009-11-23 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Nocturia
MeSH Terms: conditions — Nocturia | interventions — darifenacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- darifenacin (Experimental)
  Interventions: Drug: darifenacin
- Sugar Pill (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: darifenacin — 7.5 or 15 mg darifenacin, once a day for 6 weeks
  Other Names: Enablex
  Arms: darifenacin
Drug: Placebo — Placebo pill, once a day, for six weeks
  Arms: Sugar Pill

SUMMARY:
The purpose of this study is to evaluate the efficacy of darifenacin in the treatment of moderate to severe nocturia in patients with overactive bladder and who do not have non-urologic causes of nocturia.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be aged 21-70, inclusive.
* Subject mush have given written, personally signed and dated informed consent.
* Subject must be diagnosed with overactive bladder.
* Subject must have a nocturia frequency of greater than or equal to 3 episodes a night.
* Subject must be male or non-pregnant, non-lactating female who agrees to comply with applicable contraceptive requirements.
* Subject understands and is able, will a nd and likely to fully comply with study procedures and restrictions.

Exclusion Criteria:

* Subject has any concurrent chronic or acute illness or unstable medical condition either treated or untreated that could confound the results of safety assessments, increase risk to the subject or lead to difficulty complying with the protocol.
* The subject has a known or suspected allergy, hypersensitivity, or other medical contraindications to darifenacin (Enablex®) (or its components).
* The subject has concomitant diseases in which the use of anticholinergic drugs is contraindicated, e.g. urinary retention, bladder obstruction, gastric retention and other severe decreased gastrointestinal motility conditions, uncontrolled narrow-angle glaucoma, myasthenia gravis, severe hepatic impairment (Child Pugh C), severe ulcerative colitis, toxic megacolon, and patients who are at risk for these conditions.
* Subject is taking another drug which is considered to have significant anticholinergic activity.
* Use of drugs known to effect cognition, alertness or drowsiness, such as benzodiazepines, sedating antihistamines, opioids, or other sedative hypnotic drugs.
* Subject has moderate to severe obstructive sleep apnea (Apnea/Hypopnea Index ≥ 15)
* Subject has a medical condition other than OAB that is the most likely cause of the subject's nocturia (e.g., primary sleep disorder, polydipsia, polyuria).
* Subject has taken another investigational drug or taken part in a clinical trial within the last 30 days prior to Screening.
* The female subject is pregnant or lactating.
* Subjects with a urine drug screen positive for stimulants, barbiturates, hallucinogens, opiates, cocaine, cannabis, or amphetamines

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-11; Study Completion 2010-07 (Estimated)